CLINICAL TRIAL: NCT05073380
Title: PROmoting Early Childhood Outside (PRO-ECO): An Outdoor Play Intervention for Children Aged 3 to 5 Years in Early Childhood Education Centres
Brief Title: PROmoting Early Childhood Outside (PRO-ECO)
Acronym: PRO-ECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Mariana Brussoni, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-03912-A001
Record Dates: First submitted 2021-09-13; First posted 2021-10-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Child Development
Keywords: Children's outdoor play; Children's outdoor risky play; Early childhood education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Outdoor play is an essential component of childhood development, including supporting children's cognitive, physical, emotional, and social growth. Currently, the YMCA early learning and child care centres (ELCCs) host children within childcare settings, with outdoor playtime governed by institutional regulations.
  Interventions: Behavioral: Wait List Group - Normal Daily Practice
- Intervention (Sham Comparator): The PRO-ECO intervention to increase the quality of outdoor play involves four primary components:
  1. Modifying YMCA GV's outdoor play policies The ELCC policy on outdoor play requirements and procedures will be modified in conjunction with YMCA management.
  2. ECE training ECEs will undergo training delivered by YMCA of Southwestern Ontario that includes the importance of outdoor risky play, along with other online training tools along with resources on supporting outdoor play. There will also be ongoing as-needed supportive training and mentorship provided by YMCA senior managers and research team, along with peer mentorship and support.
  3. ELCC outdoor space modification This includes designing and implementing tailored modifications for each centre's outdoor play space developed by landscape architecture students.
  4. Parent engagement We will host parent-engagement events and opportunities to increase knowledge of the importance of outdoor play.
  Interventions: Behavioral: Intervention Group - PRO-ECO Intervention

INTERVENTIONS:
Behavioral: Intervention Group - PRO-ECO Intervention — The PRO-ECO intervention will be tailored to individual sites. Through collection of focus group and baseline data, the intervention will be further refined to provide site-specific adjustments, such as specific materials in the built environment design modification or targeted training. Identified features of effective interventions outlined in the literature have informed the development of the intervention foundation and potential tailoring.
  Arms: Intervention
Behavioral: Wait List Group - Normal Daily Practice — ELCCs that are randomly assigned to the waitlist group will participate in their normal daily practice, including standard curriculum and outdoor play time. Once post-data collection is complete, wait list sites will be given the PRO-ECO intervention.
  Arms: Control

SUMMARY:
Licensed early learning and childcare centres (ELCCs) can provide children with rich opportunities for outdoor play that they may not otherwise experience in their home or community. However, many ELCCs struggle to provide high quality and stimulating outdoor play time. The primary aim of our study is to develop, implement and test a comprehensive multi-component intervention, the PROmoting Early Childhood Outside (PRO-ECO), to build capacity for, and address the complexities of building support for outdoor play in early childcare centre settings. This is to ultimately increase children's access to engaging outdoor spaces for play.

Our overarching goal is to develop and evaluate a comprehensive multi-component intervention, called the PROmoting Early Childhood Outside (PRO-ECO). This intervention is to increase children's outdoor play and the diversity of outdoor play behaviour in Canadian ELCC settings providing full-day licensed care for preschoolers. The PRO-ECO integrates development of policies and procedure, early childhood educator (ECE) training and mentorship, outdoor space modifications and, parent/caregiver engagement.

The PRO-ECO intervention will be co-developed, implemented and evaluated in partnership with the YMCA of Greater Vancouver (YMCAGV). A wait-list control cluster randomised trial design (RCT) will evaluate the effectiveness of the intervention and how it can be modified to tackle barriers in diverse settings.

DETAILED DESCRIPTION:
The design of this study is a pilot wait-list control cluster randomised trial (RCT) with two arms. The two arms consist of 1) a PRO-ECO intervention group and 2) a wait-list control group. A mixed-methods approach will be used to collect qualitative and quantitative data designed to meet the study objectives. Quantitative data collection will support evaluation of the primary outcome variables and qualitative data will be collected to assess the acceptability, effectiveness, and feasibility of the implementation of the intervention. Qualitative data will be collected concurrently with quantitative data and will allow researchers to explore how participants experience the intervention.

Participant inclusion and exclusion criteria is divided into three distinct sets of levels- 1) organization level, 2) adult individual participation, and 3) child participation.

1. Organization level Inclusion criteria of the ELCCs include approving participation in this study. Following this, sites will be selected based on geographic area and demographics of neighbourhood served, physical characteristics of the ELCC outdoor space (e.g., size, at grade or not), readiness of program (as assessed by YMCA senior staff), and time spent participating in outdoor play. These variables will be measured based on a pretrial inventory and infrastructure survey, and census subdivision. ELCCs that do not meet the inclusion characteristics based on these measurements may be excluded.
2. Adult individual participation Inclusion criteria for adult participants include being ECEs or staff (administrators, directors, and supervisors) at the participating YMCAGV ELCCs that provide full day childcare for preschool children.
3. Child individual participation Inclusion criteria for child participation includes being between the ages of 2.5-6 years, currently enrolled in one of the participating YMCAGV ELCCs, and obtaining parental consent for their participation in the study. Children will be excluded from the measurement portion of the study if their parent does not provide informed consent, however, all children attending the program will be exposed to the intervention.

The RCT will be conducted in 8 ELCCs operated by the YMCA GV. Individual ELCCs will serve as the unit of randomization, with 4 intervention sites and 4 wait-list control sites composing the final sample. Intervention sites will receive the intervention immediately following baseline data collection, whereas wait-list control sites will receive the intervention 6 months later. Data on outcome measures will be collected at three time points- 1) Time 1 - Baseline, prior to intervention implementation, 2) Time 2 - 6-month follow-up (4 months following implementation of the intervention within the intervention group, and 3) Time 3 - 12-month follow-up (10 months post-intervention for intervention group, 4 months post-intervention for the wait-list control group). Thus, outcome data will assess short-term and long-term outcomes within the intervention group and short-term outcomes within the wait-list control group. Baseline and post-intervention data will be included in the analysis, controlling for the cluster design.

Baseline and post-intervention data collection will occur during the Fall and Spring seasons to ensure similar weather patterns at all time points, which in Metro Vancouver involves extensive rain fall, as weather has been shown to impact outdoor play time.

As per study inclusion criteria, study participants will include children aged 2.5-6 years at 8 selected YMCA GV sites. This also includes the engagement of ECEs, supervisors, and managers. Parents of children will also be invited to participate in focus groups, consent provision, and information sharing. ELCCs will appoint a staff research lead to work closely with the research team on all phases of the project. Recruitment of children and parents will occur through the staff research lead at each ELCC. Letters and/or emails home and face-to-face conversations will promote recruitment. The research team will be actively involved with staff at each site to ensure they are provided information and direction on participant recruitment policies and procedures. The staff research lead at each ELCC will administer consent forms to families.

We will inform parents/caregivers of children enrolled in the participating YMCA GV ELCCs about our study in various ways within the YMCA GV organization. This includes via online communications and info sessions. Adult participants for the qualitative focus group be recruited internally through the YMCA GV. When contacted by prospective participants including ECEs and staff, we will provide details of the study through phone or via email. On the interview day, the consent and the overall interview procedure will be further explained to participants. The focus groups will be conducted through Zoom. Once procedures are explained and consent reviewed, we will invite participants to sign the consent forms and complete the demographic survey, and email scanned copies to the UBC research team.

For the primary outcome, proportion of play occurrence, in comparison to non-play occurrence, child play behaviours will be assessed utilizing observational behaviour mapping methods. To conduct observational behaviour mapping, two research staff will be on site at each of the 8 ELCCs to collect pre-determined data related to play behaviour during outdoor free play. Behaviour mapping assessments will be performed through scanning identified quadrants throughout the outdoor play space. Simultaneous to the in-situ coding, the research staff will be taking video recordings of the quadrants they are observing. Videos will be coded at 15-second intervals for play type, including functional play, play with rules, imaginative play, constructive play, exploratory play, restorative play, and non-play. The proportion of play occurrence (vs. non-play occurrence) will be summarized by treatment group using frequency and percentages. We will compare proportions at baseline and follow-ups.

The diversity of children's play behavior when participating in outdoor play is a secondary outcome, and will be coded in situ and via review of the videos. We will compare the diversity of types of play occurring at baseline and follow-up by comparing proportions of the various play types, including physical play, expressive play, play with rules, imaginative play, exploratory play, restorative play, bio play, digital play and non-play.

ECEs' attitudes toward outdoor risky play is a secondary outcome, and will be assessed using the Teacher Tolerance of Risk in Play Scale (T-TRiPS).

The quality of outdoor spaces will be an additional outcome. The Seven Cs audit tool will form the basis for the assessment of quality of outdoor space at all early childhood education centre sites, guide development of the plan for modification of the outdoor environment, and to reassess at intervention early childhood education centre sites after implementation of the PRO-ECO intervention.

The same procedures described above will be followed to collect post-intervention data. We will also collect ECEs and staff's acceptability of the PRO-ECO intervention. This will be done utilizing a combination of focus group discussion and administrative data.

ELIGIBILITY:
Participant inclusion and exclusion criteria is divided into three distinct sets of levels- 1) organization level, 2) adult individual participation, and 3) child participation.

1. The YMCAGV ELCC site inclusion criteria:

   We will select ELCCs providing full day care to preschool children to include in the study in consideration of different variables - geographic area and demographics of neighbourhood served, physical characteristics of the ELCC outdoor space (e.g., size, at grade or not), readiness of program (as assessed by YMCA senior staff), and time spent participating in outdoor play. These variables will be further explored with the YMCA GV to determine priority site inclusion criteria and finalize site selection.
2. Adult participation inclusion criteria:

   -Being early childhood educators (ECEs) or staff (e.g., administrators, directors and supervisors) at the participating YMCA GV ELCCs.
3. Child participation inclusion criteria:

   * Being between the ages of 2.5 to 6 years;
   * Currently enrolled in one of the participating YMCAGV ELCCs;
   * Obtained parental consent for their participation in the study.

Ages: 30 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Assessing child participation in outdoor free play by identifying prevalence of play | Intervention Group - Change of prevalence of play at 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Change of prevalence of play at 5-months post-intervention (Fall 2022)
  To assess children's participation in outdoor free play at ELCCs, an observational behavior mapping (OBM) methodology will be used. OBM involves understanding how an environment supports movement through mapping, recording, and analyzing geographically located data.
  OBM involves trained research assistants taking observations at the 8 participating YMCA sites as children participate in designated outdoor playtime. OBM assessments will be performed by scanning designated observational zones throughout the outdoor play space. The observational data will be collected based on the 'space' of the ELCC, not by individual child. If there is no child in an observational zone, there will be no data collected at that point. Within each observational zone, children's play activities will be coded in 15-second increments.
  For the primary outcome measure, the categories being collected are 'play' (child observed for that data point is engaged in play) and 'non-play' (child is not playing).

SECONDARY OUTCOMES:
Assessing the diversity of play types children engage in | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  In addition to assessing time spent participating in outdoor free play, further detail on the type of play behaviour and movement is important to understanding children's outdoor free play in ELCC settings. OBM as described above will be used to assess the diversity of outdoor free play through 'play type'. Play types to be coded include physical play, expressive play, play with rules, imaginative play, exploratory play, restorative play, bio play, digital play and non-play.
Quality of early childhood education centres' outdoor play spaces | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  The Seven Cs assessment tool, designed to provide guidance in the design of outdoor play spaces for children in early childhood settings, is based on seven criteria- character, context, connectivity, change, chance, clarity, and challenge. The Seven Cs will form the basis for the assessment and re-assessment of the quality of outdoor space at all centres, and will guide development of the plan for modification of the outdoor environment.
Early childhood educators' attitudes towards outdoor risky play | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  The effect of the PRO-ECO intervention on early childhood educators' tolerance of risk in play will be assessed utilized the Teacher Tolerance of Risk in Play Scale; validated for use as a measure of intervention effects aimed at increasing children's access to risky play.
Acceptability and feasibility of PRO-ECO intervention | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  Qualitative data, including focus groups and/or individual key informant interviews, will be conducted with early childhood educators, early childhood education centre administrators, and parents respectively. To facilitate discussion, examples of pedagogical narration will be included- this will assist with discussions on how the intervention influenced the children and their outdoor play, as well as the groups' personal experiences with the intervention.
Economic analysis of PRO-ECO intervention | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  An economic evaluation will examine the costs of implementation of the intervention, as well as the potential benefits. YMCA administrative data will be abstracted to collect early childhood educator turnover, children's attendance rates, and reported incidents of challenging child behaviors.

OTHER OUTCOMES:
Children's psychosocial strengths | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  The Strengths and Difficulties Questionnaire teacher version will be utilized to assess the psychosocial strengths of children, including emotional symptoms, conduct problems, hyperactivity and inattention, peer relationship problems, and prosocial behaviour.
Children's relationship to outdoor play | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  Children's confidence, motivation, knowledge, and understanding of outdoor free play will be captured through the Early Childhood Educator's pedagogical narratives, focus groups, and interviews.
Child health | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  Child health will be measured through injury incidents, abstracted through early childhood education centres' incident report forms.
Child well-being | Intervention Group - Baseline (Fall 2021), 5-months/10-months post-intervention (Spring 2022/Fall 2022); Wait List Control Group - Baseline/post-baseline (Fall 2021/Spring 2022), 5-months post-intervention (Fall 2022)
  The Preschool Social Behaviour Scale- Teacher form, as well as the Strengths and Difficulties Questionnaire teacher version will be used to measure types of aggression and emotional symptoms respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Brussoni, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data set will be available from Dr. Brussoni upon reasonable requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting upon publication of the RCT results until five years after publication.
Access Criteria: Dr. Brussoni will review requests and share supporting information as indicated above with researchers and students going similar research interests.

REFERENCES:
- [Derived] Ramsden R, Han CS, Mount D, Loebach J, Cox A, Herrington S, Bundy A, Fyfe-Johnson A, Sandseter EBH, Stone M, Tremblay MS, Brussoni M. An Intervention to Increase Outdoor Play in Early Childhood Education Centers (PROmoting Early Childhood Outside): Protocol for a Pilot Wait-list Control Cluster Randomized Trial. JMIR Res Protoc. 2022 Jul 12;11(7):e38365. doi: 10.2196/38365. PMID 35819829